CLINICAL TRIAL: NCT00248924
Title: Outcomes Of Social Service Programs For Homebound Older Adults
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The New York Community Trust (Other)
Responsible Party: Mary E. Charlson, Weill Cornell Medical College
Other Study IDs: 0101-561
Record Dates: First submitted 2005-09-13; First posted 2005-11-04 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Homebound; Elderly
Keywords: Social service intervention; Social support; Elderly; Homebound; Quality of life
MeSH Terms: interventions — Social Work

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Social Services

SUMMARY:
The objective of this prospective study is to document the impact of social service interventions (including meals, telephone reassurance, and friendly visiting)provided by the Burden Center, a model community social service agency, on overall quality of life.

DETAILED DESCRIPTION:
Specific outcomes include mental and physical function as measured by the SF-36, and depressive symptoms as measured by the CES-D depression scale. The hypothesis is that a multicomponent social service intervention program that provides social support and reduces social isolation can prevent depression and decline in quality of life in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* All new clients of the Burden Center for the Aging who are homebound, out of the home less than one time per week, and cognitively intact will be eligible for enrollment.

Exclusion Criteria:

* Clients unable to give informed consent such as those suffering from a major psychiatric disease or those who are not cognitively able to give informed consent will be excluded.
* Clients who refuse to participate will be excluded

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2001-04; Study Completion 2003-02

PRIMARY OUTCOMES:
Quality of life Depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

REFERENCES:
- [Background] Charlson ME, Peterson JC, Syat BL, Briggs WM, Kline R, Dodd M, Murad V, Dionne W. Outcomes of community-based social service interventions in homebound elders. Int J Geriatr Psychiatry. 2008 Apr;23(4):427-32. doi: 10.1002/gps.1898. PMID 17918183